CLINICAL TRIAL: NCT01322477
Title: Contribution of F-18 Fluoro-Deoxy-Glucose PET/CT (Positron Emission Tomography) to the Assessment of HCC (Hepato-cellular Carcinoma) Treatment Efficiency
Acronym: HCC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Other Study IDs: 0022-11-HMO
Record Dates: First submitted 2011-02-14; First posted 2011-03-24 (Estimated); Last update posted 2011-03-24 (Estimated); Status verified 2011-01

CONDITIONS: Hepatocellular Carcinoma
Keywords: Identification of treatment efficacy in patients with advanced HCC by PET/CT F18-FDG
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Hepatocellular Carcinoma: Patients with advanced HCC
  Interventions: Other: F18-FDG PET/CT

INTERVENTIONS:
Other: F18-FDG PET/CT

SUMMARY:
HCC (Hepato-cellular Carcinoma) is the fifth most frequent cancer in humans and its prevalence is growing. The most effective treatment of HCC is surgical and includes resection and liver transplantation; however, only 20% of the patients can be treated surgically. Local interventional therapy, such as radiofrequency (RF) ablation and transarterial embolization is also used.

Recurrence rate is very high, and extrahepatic disease develops in about 30% of the cases and in up to 20% after liver transplantation.

Systemic treatment is thus an option. Sorafenib (multi-kinase inhibitor) is the first agent to significantly improve the overall survival in advanced HCC. However, the drug has serious side effects and is very expensive.

PET/CT with F18-FDG is a common tool for systemic evaluation and staging of various tumors.

The value of the FDG PET for evaluation of HCC is controversial, in particular due to the unique metabolic pathway of glucose in the HCC cells. Since 2007 more and more studies suggest the feasibility of FDG PET/CT for monitoring local recurrence (especially after RF) and metastatic spread of HCC, including detection of active disease only suspected by AFP (alphafoetoprotein) elevation.

Early detection of treatment response to therapy by whole body FDG PET/CT allows for change of treatment as early as possible,when the tumor is non-responsive before serious side effects appear or before depletion of body resources.

The aim of our study is to investigate the contribution of FDG PET/CT to assessment of treatment response.

ELIGIBILITY:
Inclusion Criteria:

* advanced HCC for systemic treatment

Exclusion Criteria:

* HCC only localized in liver,
* Other liver disease (e.g. metastases and benign lesions)

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Advanced HCC
Sampling Method: Non-Probability Sample
Enrollment: 25

PRIMARY OUTCOMES:
Measure of extent and intensity (standardized uptake value - SUV) of disease demonstrated on PET/CT images before and after treatment. | 12 weeks: PET/CT performed before treatment and every 4 weeks, after end of each treatment twice
  On each PET/CT study diseased tumor activity in the liver and extra-hepatic tissue will be localized and measured on the CT part of the scan (at least two maximal length values), and on the PET part of the scan SUV max value will be calculated by the machine software. Visual appreciation will also be noted.

SECONDARY OUTCOMES:
Prediction of treatment efficiency | 12 weeks
  Comparison between clinical outcome and PET/CT dynamic changes, measured as explained above.

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Hebrew University Medical Center, Jerusalem, Israel